CLINICAL TRIAL: NCT00776854
Title: Noveon Laser Treatment to Effect Bioburden Reduction or Elimination in Diabetic Foot Ulcer: A Davice Performance Clinical Study
Brief Title: Bioburden Reduction of Diabetic Foot Ulcer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nomir Medical Technologies (Industry)
Responsible Party: Alan Robbin, M.D., Nomir Medical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12.001a
Record Dates: First submitted 2008-10-18; First posted 2008-10-21 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

INTERVENTIONS:
Device: Noveon laser — 870 and 930nm wavelengths

SUMMARY:
Study to see if a laser can get rid of bacateria called MRSA in your diabetic ulcer

ELIGIBILITY:
Inclusion Criteria:

* 18 and older
* Diabetic foot ulcer
* MRSA positive

Exclusion Criteria:osteomylelitis pregnancy allery to e mycin

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-07 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Decrease of Bioburden Effect In diabetic Foot Ulcer | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nomir Medical, Waltham, Massachusetts, United States